CLINICAL TRIAL: NCT06687785
Title: A Comparison of the Clinical and Radiographic Results of the Entire Papilla Preservation (EPP) Technique and Conventional Flap Surgery (CFS) Technique in the Treatment of Isolated Intrabony Defects at 6 Months
Brief Title: Entire Papilla Preservation and Conventional Flap Surgery in Treating Intrabony Defects: A 6-Month Clinical Trial
Status: Active, not recruiting | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Fatma Uçan Yarkaç, Associate Professor, Dr., Necmettin Erbakan University
Other Study IDs: 20576
Record Dates: First submitted 2024-11-07; First posted 2024-11-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Periodontal Intrabony Defect
Keywords: intrabony defect; conventional flap surgery; bone graft; entire papilla preservation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Entire Papilla Preservation Technique: The Entire Papilla Preservation Technique (EPP) is a novel surgical approach aimed at enhancing periodontal regeneration, particularly in the treatment of deep intrabony defects. This technique is characterized by its focus on preserving the entire interdental papilla, which is crucial for both functional and aesthetic outcomes in periodontal therapy. The EPP technique involves creating a tunnel-like undermining incision that allows access to the defect while maintaining the integrity of the papilla, thereby minimizing trauma to the surrounding soft tissues
  Interventions: Procedure: Entire Papilla Preservation Technique
- Conventional Flap Surgery: In periodontology, the traditional flap surgery technique is a well-established surgical approach used for the treatment of periodontal diseases, especially in cases with deep periodontal pockets. This technique involves the lifting of a mucoperiosteal flap in the buccal and lingual direction to gain access to the underlying periodontal tissues and allows for thorough debridement of root surfaces and removal of diseased tissue.
  Interventions: Procedure: Conventional Flap Surgery Technique

INTERVENTIONS:
Procedure: Entire Papilla Preservation Technique — A buccal intrasulcular incision was made in the tooth with the defect and a vertical incision was made extending from the buccal center of the tooth to the mesial papillary crest and crossing the mucogingival line. Then, using a micro periosteal elevator, a full-thickness mucoperiosteal flap was lifted from the incision site to the defect under the papilla. After removal of the granulation tissues in the area, bone graft was applied for regenerative purposes and the vertical incision was sutured with 6/0 polypropylene suture using simple suture technique.
  Other Names: EPP
  Groups: Entire Papilla Preservation Technique
Procedure: Conventional Flap Surgery Technique — After buccal and lingual intrasulcular incisions were made to eliminate the teeth and papillae adjacent to the defect, a full-thickness mucoperiosteal flap was raised in the vestibular and lingual direction with a periosteal elevator. After removal of the granulation tissues in the area, bone graft was applied for regenerative purposes and the papillary incisions were sutured with 5/0 polypropylene suture using simple suture technique.
  Other Names: CFS
  Groups: Conventional Flap Surgery

SUMMARY:
Intraosseous defects are characterized by vertical bone loss within the borders of the alveolar bone surrounding the teeth due to periodontal disease and are considered a clinically concerning condition. Treatment of intraosseous defects involves regenerative techniques aimed at reconstructing lost periodontal structures (including bone, cementum and periodontal ligament). In the process of periodontal regeneration, it is of great importance that the blood clot attached to the root surface is protected from mechanical and microbiological factors and remains in a stable biological environment. Post-surgical wound dehiscence can lead to impaired clot stabilization and infection, negatively affecting the healing process and thus jeopardizing the results of the treatment.

Regenerative therapies using conventional flap surgery have been reported to provide significant improvements in clinical attachment levels, but carry a high risk of loss of attachment if flap management is inadequate. Furthermore, complications such as difficulty in primary closure, risk of membrane exposure and tissue detachment have been observed with conventional flap techniques. Various minimally invasive flap surgery techniques have been developed to prevent these complications. One of the minimally invasive periodontal flap techniques is the full papillary preservation technique. Unlike traditional methods, this innovative approach provides vertical access to the defect area from the buccal and lingual adjacent areas without any incision in the papillary region. This technique reduces the risk of wound healing failure and exposure of regenerative biomaterials due to the fully preserved interdental papilla over the bony defect. The aim of our study is to compare the short-term (6 months) radiographic and clinical results of the Entire Papilla Preservation (EPP) technique with the Conventional Flap Surgery (CFS) technique.

ELIGIBILITY:
Inclusion Criteria:

* Systemic health
* Probing depth (PD) ≥7 mm
* Clinical attachment level (CAL) ≥7 mm
* Presence of an isolated two or three walled intraosseous defect with an intraosseous component of at least 4 mm predominantly involving the interproximal region of the affected tooth
* Full mouth plaque score (FMPS) and full mouth bleeding score ≤20%

Exclusion Criteria:

* Current smoking habit
* Presence of uncontrolled systemic diseases that prevent periodontal surgery
* Use of drugs that affect periodontal tissues
* Pregnancy and breastfeeding
* Single-walled intraosseous defects
* Defects involving the buccal and/or lingual areas of the tooth
* Inadequate endodontic treatment and/or restorations on teeth in the defect area.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Periodontitis patients with isolated intrabony defects
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Probing Depth | 6 MONTH
  Probing Depth (PD) refers to the distance from the gingival margin to the base of the periodontal pocket. It is expressed in mm and a high measurement is a clinically unfavorable value.
Clinical Attachment Level | 6 MONTH
  Clinical Attachment Level (CAL) is defined as the distance from the cementoenamel junction (CEJ) to the base of the periodontal pocket. It is expressed in mm and a high measurement is a clinically unfavorable value.
Gingival Recession | 6 MONTH
  Gingival Recession (GR) refers to the apical migration of the gingival margin, resulting in exposure of the root surface. While it should be 0 in healthy individuals, an increase is a bad value.

SECONDARY OUTCOMES:
Visual analogue scale | for 2 weeks after treatment
  Postoperative patients were asked to fill out a visual analogue scale to determine their pain levels on the 1st, 3rd, 7th and 14th days. This scale was scored between 0-100, with 0 indicating no pain and 100 indicating unbearable pain.
Early healing index. | 1 week after treatment
  The healing status in the first postoperative week was evaluated with a score between 1(perfect healing) and 5(worst healing) using the early healing index.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma UCAN YARKAC, assoc. prof., Principal Investigator — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Faculty of Dentistry, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stavropoulos A, Karring T. Five-year results of guided tissue regeneration in combination with deproteinized bovine bone (Bio-Oss) in the treatment of intrabony periodontal defects: a case series report. Clin Oral Investig. 2005 Dec;9(4):271-7. doi: 10.1007/s00784-005-0002-7. Epub 2005 Jul 12. PMID 16010581
- [Result] Aslan S, Buduneli N, Cortellini P. Entire Papilla Preservation Technique: A Novel Surgical Approach for Regenerative Treatment of Deep and Wide Intrabony Defects. Int J Periodontics Restorative Dent. 2017 Mar/Apr;37(2):227-233. doi: 10.11607/prd.2584. PMID 28196163
- [Derived] Yarkac FU, Yildiz K, Kalender ME, Ogutcen O. Clinical and radiographic outcomes of entire papilla preservation versus open flap debridement using bovine-derived xenograft and leukocyte- and platelet-rich fibrin in the treatment of isolated intrabony defects. BMC Oral Health. 2025 Oct 21;25(1):1639. doi: 10.1186/s12903-025-07008-9. PMID 41121124